CLINICAL TRIAL: NCT06040411
Title: The Effect of Acupressure on Preoperative Anxiety and Postoperative Pain and Nausea-Vomiting in ENT Surgery
Brief Title: The Effect of Acupressure on Preoperative Anxiety and Postoperative Pain and Nausea-Vomiting
Acronym: Acupress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Tugba CAM YANIK, Principal Investigator Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mersin University.
Record Dates: First submitted 2023-08-22; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Anxiety State; Pain; Vomiting; Nausea
Keywords: pain; ENT patients
MeSH Terms: conditions — Anxiety Disorders; Pain; Vomiting; Nausea | interventions — Acupressure

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: The statistician was blinded to analyze the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (experimental) (Experimental): The order of application was determined by lottery. HT7, LI4 and EX-HN3 points were applied respectively. Before starting the application, the area around to be pressurized was gently rubbed with the palm of the hand for 20-30 seconds. The surrounding tissue was relieved by rubbing gently. After rubbing, pressure was applied to the point determined based on the pain threshold level of each individual with a depth of 1-1.5 cm with the thumb for 5 seconds, rested for 2 seconds and the application was continued for 2 minutes. Acupressure was applied to each point for 2 minutes and the total application time was 15 minutes on average (for 5 points).
  Interventions: Other: Acupressure
- Standard of care (No Intervention): Standard care was given.

INTERVENTIONS:
Other: Acupressure — Acupressure was applied to each point for 2 minutes and the total application time was 15 minutes on average (for 5 points). During the application, the most appropriate position in which the individual would be comfortable was preferred, taking into account the privacy of the individual. First of all, the supine position was preferred, and alternatively, the sitting position was preferred. At the end of the application, it was ensured that the person was in a position that he/she was comfortable.
  Other Names: Acupress
  Arms: Study Group (experimental)

SUMMARY:
The study was conducted in the ENT Clinic of Mersin Şehir Training and Research Hospital between June 1 and December 1, 2021, with a total of 60 adult patients, 30 in the study group and 30 in the control group, who met the inclusion and exclusion criteria.

DETAILED DESCRIPTION:
In the study, 60 patients were randomly assigned to the study and control groups. The study group (n = 30) included Shen Men, the 7th acupuncture point (HT7) of the heart meridian located between the ulna and pisiform bones on the radial side of the flexor carpi ulnaris tendon, EX-HN3 (Yintang) located in the middle of the beginning of both eyebrows and the thumb and the LI4 points located in the space between the index finger (between the 1st and 2nd metacarpal bones of the hand, in the middle of the 2nd metacarpal bone on the radial side) were applied for an average of 15 minutes. No intervention didn't made to the control group (n = 30). The primary outcome of the study is the effect of acupressure on the state and trait anxiety level of patients. The secondary outcome of the study is the effect of acupressure on pain and nausea and vomiting level in patients. Anxiety levels of the patients were evaluated before and 15 minutes after acupressure application; pain levels were evaluated at the 4th postoperative hour, before going to bed at night (22.00), waking up in the morning (08.00) and at discharge; nausea and vomiting levels were evaluated in the first 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Emergency ENT surgery,
* Refused to participate in the research,
* Did not sign the Informed Consent Form,
* Have a physical problem that prevents the application of acupressure to EX-HN3 (Yintang), LI4 and HT7 points,
* Diagnosed with anxiety, panic attacks and taking medication for anxiety,
* Previous surgical experience,
* Under 18 and over 65,
* People with vision, hearing and perception problems,
* unable to read and write Turkish,
* Have any problem that prevents them from communicating cognitively, emotionally and verbally,
* Experience in acupressure,
* Patients who have received sedative medication before surgical intervention didn't be included in the study.

Exclusion Criteria:

* Emergency ENT surgery,
* Refused to participate in the research,
* Did not sign the Informed Consent Form,
* Diagnosed with anxiety, panic attacks and taking medication for anxiety,
* Previous surgical experience
* Under 18 and over 65,
* People with vision, hearing and perception problems,
* unable to read and write Turkish,
* Have any problem that prevents them from communicating cognitively, emotionally and verbally,
* Experience in acupressure,
* Patients who have received sedative medication before surgical intervention didn't be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Anxiety evaluated using the State Anxiety Scale | Change from before implementation and immediately after, 15th minutes after implementation
  Scores ranging from 20 to 80 points are obtained in the scale. In the total score obtained from the scale in scoring the scale, 0-19 points indicate the absence of anxiety, 20-39 points indicate mild anxiety, 40-59 points indicate moderate anxiety, and 60-79 points indicate severe anxiety level. Higher state anxiety scores indicate that anxiety level is also high

SECONDARY OUTCOMES:
Numerical Pain Scale | Change from the 4th hour after surgery, through the discharge, an average of 2 days
  In this scale, the patient is asked to describe the severity of his/her pain in numbers, and the scale consists of a horizontal line, with "0" or "no pain" at the starting point and "10" or "unbearable pain" at the end point. The numbers from 0 to 10 are equally spaced on the horizontal line and 1-3 is defined as mild pain, 4-6 as moderate pain and 7-10 as severe pain.
Nausea and vomiting | Change from surgery to the first 24 hours
  The responses for each item are scored between zero (least discomfort) and four (most discomfort). The scores obtained from the eight items are summed to obtain a total score. The maximum score that can be obtained from the index is 32, which is also considered as the most severe symptom occurrence experience score.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay ALTUN UĞRAŞ, PhD, Study Director — Mersin University; Serpil YÜKSEL, PhD, Principal Investigator — Necmettin Erbakan University; Bahar TAŞDELEN, PhD, Principal Investigator — Mersin University; Seda TÜRKİLİ, Doctor, Principal Investigator — Mersin City Hospital; Serkan TÜRKİLİ, Doctor, Principal Investigator — Mersin City Hospital; Ahmet KARAMAN, PhD, Principal Investigator — Mersin University
Locations (1):
- Tuğba ÇAM YANIK, Yenişehir, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No